CLINICAL TRIAL: NCT01117428
Title: An Open-label, Multi-center Phase I Dose Escalation Study to Investigate the Safety and Tolerability of Multiple Doses of Sym004 in Patients With Advanced Solid Tumors
Brief Title: Sym004 in Patients With Advanced Solid Tumors
Status: Completed | Phase: Phase 1 / Phase 2 | Type: Interventional
Sponsor: Symphogen A/S (Industry)
Responsible Party: Sponsor
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: Sym004-01; 2009-017119-13 (EudraCT Number)
Record Dates: First submitted 2010-04-23; First posted 2010-05-05 (Estimated); Results first posted 2017-07-12 (Actual); Last update posted 2018-10-15 (Actual); Status verified 2018-09

CONDITIONS: Metastatic Colorectal Cancer
Keywords: Advanced solid tumors; Metastatic colorectal Cancer
MeSH Terms: conditions — Colorectal Neoplasms | interventions — futuximab

STUDY DESIGN:
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: Yes | FDA-regulated Device: No

ARMS (1):
- Sym004 (Experimental)
  Interventions: Drug: Sym004

INTERVENTIONS:
Drug: Sym004 — In part A, patients in all dose cohorts will continue weekly treatment with the assigned dose of Sym004 until disease progression.
  In Part B, patients will continue weekly treatment with the tolerated dose of Sym004 until disease progression.
  In Part C, patients will receive weekly doses of Sym004 at the dose level below 12 mg/kg i.e. 9 mg/kg until disease progression.
  In Part D and E, patients will receive doses of Sym004 administered every 2 weeks at dose level 12 mg/kg and 18 mg/kg, respectively until disease progression.
  In Part F, patients will receive a single loading dose of 9 mg/kg followed by weekly doses of 6 mg/kg.

SUMMARY:
This trial is designed as a multi-centre, open label, dose-escalation, phase I trial and consists of five parts.

DETAILED DESCRIPTION:
Part A investigates the safety and pharmacokinetics (PK) of escalating weekly dosing of Sym004 in patients with recurrent advanced solid tumors.

Part B and C validates the safety, PK and efficacy of weekly dosing of Sym004 at the maximum tolerated dose (MTD) in a homogenous patient population with advanced metastatic colorectal cancer (mCRC) and wild-type Kirsten rat sarcoma (KRAS). Part B will be initiated when a safe dose has been established in Part A.

If MTD equals 12 mg/kg, then part C will explore the 9 mg/kg level.

Part D and E is to validate the safety, PK and efficacy when administered every 2 weeks at doses of 12 mg/kg and 18 mg/kg, respectively.

Part F is to validate safety, PK and efficacy when administered with a single loading dose of 9 mg/kg followed by weekly doses of 6 mg/kg.

ELIGIBILITY:
Inclusion Criteria:

Part A:

1. Patients with refractory or recurrent advanced late stage solid tumors without available therapeutic options .

Part B, C, D, E and F:

1. Patients with refractory or recurrent advanced mCRC and wild-type KRAS who have progressed on epidermal growth factor receptor (EGFR) Ab treatment.
2. Patients wit confirmed response while on treatment anti-EGFR Ab treatment.
3. Documented disease progression during or within 6 months after cessation of anti-EGFR Ab treatment.
4. Patients must be willing to have a biopsy performed from a tumor lesion at screening and at Visit 6.

Part A, B, C, D, E and F:

1. Histologically or cytologically confirmed diagnosis of cancer
2. Failure and/or intolerance to standard chemotherapy
3. Life expectancy of at least 3 months
4. Eastern Cooperative Oncology Group (ECOG) performance status ≤2

Exclusion Criteria:

1. Patients with clinically symptomatic brain metastases.
2. Received the following treatments prior to Visit 2:

   * Cytotoxic or cytostatic anti-cancer chemotherapy within 4 weeks
   * Total resection or irradiation of the target lesion
   * Antibody therapy within 4 weeks and vaccines within 12 weeks
   * Tyrosin kinase inhibitors within 4 weeks
   * Any investigational agent within 4 weeks
3. Diarrhea CTCAE >1
4. Skin rash CTCAE >1
5. Abnormal organ or bone marrow function.
6. Use of immunosuppressive agents for the past 4 weeks prior to trial start, including systemic corticosteroids used at doses above 20mg/day of prednisolone or equivalent.
7. History of other malignancy within 5 years prior to trial start, with the exception of basal cell carcinoma of the skin and carcinoma in situ of the cervix (not in Part A).
8. Active severe infection, any other concurrent disease or medical conditions that are deemed to interfere with the conduct of the trial as judged by the investigator.
9. Known HIV positive
10. Known active hepatitis B or C
11. Patients with known uncontrolled allergic conditions or allergy to the study drug and/or their components.
12. Clinically significant cardiac disease including unstable angina, acute myocardial infarction within six months from Visit 1, congestive heart failure, and arrhythmia requiring therapy, with the exception of extra systoles or minor conduction abnormalities and controlled and well treated chronic atrial fibrillation.
13. Significant concurrent, uncontrolled medical condition evaluated by the investigator to interfere with effect of the trial drug.

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 111 (Actual)
Dates: Start 2010-03 (Actual); Primary Completion 2015-02 (Actual); Study Completion 2015-05 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Josep Tabernero, MD, PhD, Principal Investigator — Vall d´Hebron University Hospital
Locations (7):
- South Texas Accelerated Research Therapeutics (START), San Antonio, Texas, United States
- Belgium (3):
  - UZ Brussel, Medische Oncologie, Brussels
  - UZ Gasthuisberg, Digestive Oncology Unit, Brussels
  - UZ Antwerp, Oncologie, Edegem
- Spain (3):
  - Medical Oncology Department, Vall d´Hebron University Hospital, Barcelona
  - Servicio de Oncología Médica, Hospital Universitario Virgen del Rocío, Seville
  - Hospital Clínico Universitario de Valencia, Valencia

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- [Derived] Dienstmann R, Patnaik A, Garcia-Carbonero R, Cervantes A, Benavent M, Rosello S, Tops BB, van der Post RS, Argiles G, Skartved NJ, Hansen UH, Hald R, Pedersen MW, Kragh M, Horak ID, Braun S, Van Cutsem E, Tolcher AW, Tabernero J. Safety and Activity of the First-in-Class Sym004 Anti-EGFR Antibody Mixture in Patients with Refractory Colorectal Cancer. Cancer Discov. 2015 Jun;5(6):598-609. doi: 10.1158/2159-8290.CD-14-1432. Epub 2015 May 11. PMID 25962717

RESULTS

PARTICIPANT FLOW:
Groups:
- Part A: Dose Escalation: Dose escalation in patients with refractory or recurrent advanced solid tumors.
  Sym004: 0.4 mg/kg, 0.75 mg/kg, 1.5 mg/kg, 3 mg/kg, 6 mg/kg, 9 mg/kg, 12 mg/kg, weekly - i.v. infusions
- Part B: Dose Expansion Cohort: Dose expansion cohort in patients with advanced anti-epidermal growth factor receptor (anti-EGFR) antibody refractory metastatic colorectal cancer (mCRC).
  Sym004: 12 mg/kg, weekly - i.v. infusions
- Part C: Dose Expansion Cohort: Dose expansion cohort in patients with advanced anti-EGFR antibody refractory mCRC.
  Sym004: 9 mg/kg, weekly - i.v. infusions
- Part D: Dose Expansion Cohort: Dose expansion cohort in patients with advanced anti-EGFR antibody refractory mCRC.
  Sym004: 12 mg/kg, once every 2 weeks - i.v. infusions
- Part E: Dose Expansion Cohort: Dose expansion cohort in patients with advanced anti-EGFR antibody refractory mCRC.
  Sym004: 18 mg/kg, once every 2 weeks - i.v. infusions
- Part F: Dose Expansion Cohort: Dose expansion cohort in patients with advanced anti-EGFR antibody refractory mCRC.
  Sym004: 9 mg/kg loading dose followed by 6 mg/kg, weekly - i.v. infusions
Period: Overall Study
Arm/Group | Part A: Dose Escalation | Part B: Dose Expansion Cohort | Part C: Dose Expansion Cohort | Part D: Dose Expansion Cohort | Part E: Dose Expansion Cohort | Part F: Dose Expansion Cohort
Started | 20 (0.4 mg/kg=1 0.75 mg/kg=1 1.5 mg/kg=3 3 mg/kg=3 6 mg/kg=3 9 mg/kg=6 12 mg/kg=3) | 29 | 13 | 12 | 17 | 20
Completed | 0 | 0 | 0 | 0 | 0 | 0
Not Completed | 20 | 29 | 13 | 12 | 17 | 20
Not completed — Lack of Efficacy | 1 | 0 | 0 | 0 | 0 | 0
Not completed — Adverse Event | 4 | 0 | 0 | 0 | 1 | 2
Not completed — Death | 0 | 1 | 2 | 0 | 0 | 1
Not completed — Physician Decision | 0 | 1 | 0 | 0 | 0 | 0
Not completed — Withdrawal by Subject | 0 | 0 | 1 | 0 | 0 | 0
Not completed — Progressive disease | 15 | 27 | 10 | 12 | 16 | 17

BASELINE CHARACTERISTICS:
Population: Part A: Dose escalation in patients with refractory or recurrent advanced solid tumors.
  Parts B, C, D, E and F: Dose expansion cohorts in patients wíth advanced anti-EGFR antibody refractory mCRC.
Groups:
- Part B: Dose Expansion Cohort: Dose expansion cohort in patients with advanced anti-EGFR antibody refractory mCRC.
  Sym004: 12 mg/kg, weekly - i.v. infusions
- Total: Total of all reporting groups
Arm/Group | Part A: Dose Escalation | Part B: Dose Expansion Cohort | Part C: Dose Expansion Cohort | Part D: Dose Expansion Cohort | Part E: Dose Expansion Cohort | Part F: Dose Expansion Cohort | Total
Number analyzed (Participants) | 20 | 29 | 13 | 12 | 17 | 20 | 111
Age, Categorical [Count of Participants; unit: Participants]
  <=18 years | 0 | 0 | 0 | 0 | 0 | 0 | 0
  Between 18 and 65 years | 11 | 16 | 4 | 5 | 10 | 11 | 57
  >=65 years | 9 | 13 | 9 | 7 | 7 | 9 | 54
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 13 | 14 | 6 | 6 | 4 | 6 | 49
  Male | 7 | 15 | 7 | 6 | 13 | 14 | 62
Ethnicity (NIH/OMB) [Count of Participants; unit: Participants]
  Hispanic or Latino | 5 | 1 | 0 | 0 | 1 | 0 | 7
  Not Hispanic or Latino | 15 | 28 | 13 | 12 | 16 | 20 | 104
  Unknown or Not Reported | 0 | 0 | 0 | 0 | 0 | 0 | 0
Region of Enrollment [Number; unit: participants]
  Belgium | 0 | 5 | 1 | 0 | 0 | 3 | 9
  United States | 11 | 0 | 0 | 0 | 0 | 0 | 11
  Spain | 9 | 24 | 12 | 12 | 17 | 17 | 91
Disease duration [Mean (Standard Deviation); unit: years] | 4.2 (2.7) | 3.6 (1.6) | 4.1 (2.7) | 2.8 (1.0) | 4.0 (2.9) | 3.8 (2.3) | NA (NA) — Total disease duration cannot be calculated because it is defined by cohort, not the total study population.

OUTCOME MEASURES:

1. Primary Outcome: Number of Participants With Adverse Events (AEs)
Description: The AEs were used as a primary endpoint. AEs were summarized using descriptive statistics and presented overall by system organ class and preferred term. The frequencies of AEs were presented including number and percentages of participants with events and the total number of events.
Time Frame: Visit 2 until first follow-up visit (up to 66 weeks)
Measure: Count of Participants; unit: Participants
Arm/Group | Part A: Dose Escalation | Part B: Dose Expansion Cohort | Part C: Dose Expansion Cohort | Part D: Dose Expansion Cohort | Part E: Dose Expansion Cohort | Part F: Dose Expansion Cohort
Number analyzed (Participants) | 20 | 29 | 13 | 12 | 17 | 20
Participants | 20 | 29 | 13 | 12 | 17 | 20

2. Secondary Outcome: Antitumor Activity
Description: Best Overall Response (OR) on the Full Analysis Set (FAS) according to Response Evaluation Criteria in Solid Tumors (RECIST) v1.1, based on central evaluation with confirmatory CT scan or MRI [Complete Response (CR): disappearance of all target lesions; Partial Response (PR): at least a 30% decrease in the sum of diameters of target lesions; Progressive Disease (PD): at least a 20% increase in the sum of diameters of target lesions; Stable Disease (SD): neither sufficient shrinkage to qualify for PR nor sufficient increase to qualify for PD; Overall Response (OR): CR + PR]. Baseline was defined as Visit 2 (pre-infusion). The outcome measure was measured from screening until PD.
Time Frame: Up to 62 weeks
Population: Data for Part A were presented only for the FAS. For Parts B to F, analyses and summaries were performed both for the FAS and for the per protocol population. The FAS was considered the primary analysis population.
Measure: Number (95% Confidence Interval); unit: percentage of participants
Groups:
- Part C: Dose Expansion Cohort: Dose expansion cohort in patients with advanced anti-EGFR antibody refractory mCRC.
  Sym004: 9 mg/kg weekly - i.v. infusions
Arm/Group | Part A: Dose Escalation | Part B: Dose Expansion Cohort | Part C: Dose Expansion Cohort | Part D: Dose Expansion Cohort | Part E: Dose Expansion Cohort | Part F: Dose Expansion Cohort
Number analyzed (Participants) | 20 | 29 | 13 | 12 | 17 | 20
percentage of participants
  Stable Disease | 45 [23.1 to 68.5] | 58.6 [38.9 to 76.5] | 46.2 [19.2 to 74.9] | 16.7 [2.1 to 48.4] | 70.6 [44.0 to 89.7] | 65 [40.8 to 84.6]
  Progressive Disease | 40 [19.1 to 63.9] | 24.1 [10.3 to 43.5] | 30.8 [9.1 to 61.4] | 75 [42.8 to 94.5] | 17.6 [3.8 to 43.4] | 30 [11.9 to 54.3]
  Partial Response | 0 [0 to 0] | 6.9 [0.8 to 22.8] | 7.7 [0.2 to 36.0] | 0 [0 to 0] | 0 [0 to 0] | 0 [0 to 0]
  Missing | 15 [3.2 to 37.9] | 6.9 [0.8 to 22.8] | 7.7 [0.2 to 36.0] | 0 [0 to 0] | 11.8 [1.5 to 36.4] | 5 [0.1 to 24.9]
  Not Evaluable | 0 [0 to 0] | 3.4 [0.1 to 17.8] | 7.7 [0.2 to 36.0] | 8.3 [0.2 to 38.5] | 0 [0 to 0] | 0 [0 to 0]
Statistical Analysis 1: Comparison: Part E: Dose Expansion Cohort vs Part F: Dose Expansion Cohort; Test type: Equivalence — Differences between Parts E and F in terms of Best Overall Response evaluated from screening until disease progression; p = 0.6645, Fisher Exact — No adjustment, 5% significance level

3. Secondary Outcome: Antitumor Activity Endpoints - Time-to-event Endpoints
Description: Median Progression Free Survival (PFS) was defined as the time interval without PD from start of first infusion until death or documented PD (i.e. at least a 20% increase in the sum of diameters of target lesions) according to RECIST v1.1. Patients who died without confirmed PD were considered as progressed. Patients who died or showed PD more than 21 days after last treatment were censored (i.e. were considered alive without progression on Day 21 after last treatment). Patients without events were censored at date of last scan or 22 days after last treatment, whichever occurred first.
  Median Overall Survival (OS) was defined as the time from start of first infusion until date of death from any cause. Patients alive at the time of the analysis or prematurely withdrawn from the trial (e.g. lost to follow-up or consent withdrawn) were censored for the OS analysis. In any case of censoring, the date of censoring was the last time point documenting survival status.
Time Frame: Up to 62 weeks
Measure: Median (95% Confidence Interval); unit: Months
Arm/Group | Part A: Dose Escalation | Part B: Dose Expansion Cohort | Part C: Dose Expansion Cohort | Part D: Dose Expansion Cohort | Part E: Dose Expansion Cohort | Part F: Dose Expansion Cohort
Number analyzed (Participants) | 20 | 29 | 13 | 12 | 17 | 20
Months
  Progression Free Survival | 3 [1.4 to 5.1] | 3.6 [1.4 to 5.1] | 3.3 [1.2 to 5.2] | 1.4 [1.2 to 1.4] | 3.3 [1.4 to 5.1] | 3.1 [1.4 to 3.6]
  Overall Survival | 7.9 [2.9 to 10.3] | 6.9 [3.8 to 10.4] | 6.2 [1.6 to 10.5] | 2.9 [1.1 to 13.5] | 6.3 [4 to 10.3] | 9.6 [5.5 to 12.6]

4. Secondary Outcome: Terminal Half-Life (T½)
Description: For Part A, the endpoint was not calculated. For Parts B, C and F, the endpoint was calculated for each patient following the first and fourth Sym004 infusions.
  For Parts D and E, the endpoint was calculated for each patient following the first and third Sym004 infusions.
  T½ was estimated using non-compartmental methods and actual time points.
  Outcome Measure Time Frame:
  Parts B, C and F (Weekly dosing): Sample collection at Visit 2 (1st dose from end of infusion, 1-, 2-, 4-, 8-, 24-, 48-hours) until 1 week post-infusion (168-hours) and at Visit 5 (4th dose from end of infusion, 1-, 2-, 4-, 8-, 24-hours) until 1 week post-infusion (168-hours).
  Parts D, E (Dosing every second week): Sample collection at Visit 2 (1st dose from end of infusion, 1-, 2-, 4-, 8-, 24-, 48-hours) to end of 3rd dose (from end of infusion, 1-, 2-, 4-, 8-, 24-hours) until 2 weeks post-infusion (336 hours).
Time Frame: See Time Frame in the Outcome Measure Description
Population: For Part A, data could not be reported as the endpoint was not calculated and no pharmacokinetics (PK) analysis set was defined. For Parts B to F, a PK analysis set was used.
Measure: Geometric Mean (Geometric Coefficient of Variation); unit: Hours
Groups:
- Part F: Dose Expansion Cohort: Dose expansion cohort in patients with advanced anti-EGFR antibody refractory mCRC.
  Sym004: 9 mg/kg loading dose followed by 6 mg/kg, weekly - i.v. infusion
Arm/Group | Part A: Dose Escalation | Part B: Dose Expansion Cohort | Part C: Dose Expansion Cohort | Part D: Dose Expansion Cohort | Part E: Dose Expansion Cohort | Part F: Dose Expansion Cohort
Number analyzed (Participants) | 0 | 17 | 6 | 12 | 16 | 20
Hours
  1st Dose |  | 74.8 (20.9) | 61.8 (20) | 65.6 (33.6) | 108 (18.9) | 66.6 (21.2)
  3rd Dose |  | 0 (0) | 0 (0) | 88.7 (41.8) | 120.7 (25.5) | 0 (0)
  4th Dose |  | 123.6 (38.9) | 120.7 (23.5) | 0 (0) | 0 (0) | 91.7 (24)

ADVERSE EVENTS:
Time Frame: The Adverse Event (AE) reporting period for non-serious AEs started at Visit 2 (first dosing visit) and lasted until the first Follow-up Visit (4 weeks following last dose) or end of trial if the patient was withdrawn from the trial without the Follow-up Visits being performed. The AE reporting period for Serious Adverse Events (SAEs) started when the patient signed the informed consent and lasted until termination of the trial.
Description: Any non-serious signs or symptoms occurring between Visit 1 and start of treatment at Visit 2 were recorded as medical history. In the survival period after end of trial, only SAEs with fatal outcome and SAEs considered related to Sym004 by the Investigator were collected.
Groups:
- Part A: Dose Escalation: Dose escalation in patients with refractory or recurrent advanced solid tumors.
  Sym004 - 0.4 mg/kg, 0.75 mg/kg, 1.5 mg/kg, 3 mg/kg, 6 mg/kg, 9 mg/kg, 12 mg/kg, weekly - i.v. infusions
- Part B: Dose Expansion Cohort: Dose expansion cohort in patients with advanced anti-EGFR antibody refractory mCRC.
  Sym004 - 12 mg/kg, weekly - i.v. infusions
- Part C: Dose Expansion Cohort: Dose expansion cohort in patients with advanced anti-EGFR antibody refractory mCRC.
  Sym004 - 9 mg/kg, weekly - i.v. infusions
- Part D: Dose Expansion Cohort: Dose expansion cohort in patients with advanced anti-EGFR antibody refractory mCRC.
  Sym004 - 12 mg/kg, once every 2 weeks - i.v. infusions
- Part E: Dose Expansion Cohort: Dose expansion cohort in patients with advanced anti-EGFR antibody refractory mCRC.
  Sym004 - 18 mg/kg, once every 2 weeks - i.v. infusions
- Part F: Dose Expansion Cohort: Dose expansion cohort in patients with advanced anti-EGFR antibody refractory mCRC.
  Sym004 - 9 mg/kg loading dose followed by 6 mg/kg, weekly - i.v. infusions
Arm/Group | Part A: Dose Escalation | Part B: Dose Expansion Cohort | Part C: Dose Expansion Cohort | Part D: Dose Expansion Cohort | Part E: Dose Expansion Cohort | Part F: Dose Expansion Cohort
All-Cause Mortality (participants affected / at risk) | 14/20 | 29/29 | 13/13 | 9/12 | 15/17 | 14/20
Serious Adverse Events (participants affected / at risk) | 10/20 | 16/29 | 10/13 | 7/12 | 6/17 | 7/20
Other Adverse Events (participants affected / at risk) | 18/20 | 29/29 | 13/13 | 12/12 | 16/17 | 20/20
SERIOUS ADVERSE EVENTS; cells are participants affected of the arm's N at risk (number of events):
Term (organ system) | Part A: Dose Escalation (N=20) | Part B: Dose Expansion Cohort (N=29) | Part C: Dose Expansion Cohort (N=13) | Part D: Dose Expansion Cohort (N=12) | Part E: Dose Expansion Cohort (N=17) | Part F: Dose Expansion Cohort (N=20)
Myocardial infarction (Cardiac disorders) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Ascites (Gastrointestinal disorders) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Constipation (Gastrointestinal disorders) | 1 (1) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0)
Pancreatic cyst (Gastrointestinal disorders) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Intestinal obstruction (Gastrointestinal disorders) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 1 (1) | 0 (0)
Subileus (Gastrointestinal disorders) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0)
Gastric hemorrhage (Gastrointestinal disorders) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0)
Asthenia (General disorders) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
General physical health deterioration (General disorders) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Performance status decreased (General disorders) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0)
Hyperbilirubinemia (Hepatobiliary disorders) | 0 (0) | 1 (1) | 1 (1) | 0 (0) | 0 (0) | 0 (0)
Cholangitis (Hepatobiliary disorders) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1)
Jaundice (Hepatobiliary disorders) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0)
Jaundice cholestatic (Hepatobiliary disorders) | 0 (0) | 0 (0) | 0 (0) | 2 (2) | 0 (0) | 0 (0)
Hypersensitivity (Immune system disorders) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Abdominal abscess (Infections and infestations) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Esophageal candidiasis (Infections and infestations) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0)
Peritonitis (Infections and infestations) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0)
Pneumonia (Infections and infestations) | 1 (1) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Sepsis (Infections and infestations) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0)
Urinary tract infection (Infections and infestations) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1)
Catheter site infection (Infections and infestations) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0)
Endocarditis (Infections and infestations) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1)
Fracture (Injury, poisoning and procedural complications) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0)
Infusion related reaction (Injury, poisoning and procedural complications) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Spinal fracture (Injury, poisoning and procedural complications) | 1 (2) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Blood bilirubin increased (Investigations) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Hypocalcemia (Metabolism and nutrition disorders) | 0 (0) | 2 (2) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Hypomagnesemia (Metabolism and nutrition disorders) | 1 (1) | 4 (4) | 0 (0) | 1 (1) | 2 (2) | 4 (4)
Hypophosphatemia (Metabolism and nutrition disorders) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Back pain (Musculoskeletal and connective tissue disorders) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Arthralgia (Musculoskeletal and connective tissue disorders) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1)
Neck pain (Musculoskeletal and connective tissue disorders) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0)
Neoplasm malignant (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 7 (7) | 9 (9) | 6 (6) | 4 (4) | 1 (1) | 2 (2)
Metastases to central nervous system (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Tumor pain (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0)
Spinal cord compression (Nervous system disorders) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Obstructive uropathy (Renal and urinary disorders) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Renal failure acute (Renal and urinary disorders) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1)
Bronchospasm (Respiratory, thoracic and mediastinal disorders) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Pulmonary embolism (Respiratory, thoracic and mediastinal disorders) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 1 (1) | 0 (0)
Dermatitis acneiform (Skin and subcutaneous tissue disorders) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Dermatosis (Skin and subcutaneous tissue disorders) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0)
Rash (Skin and subcutaneous tissue disorders) | 1 (1) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Shock (Vascular disorders) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Hypovolemic shock (Vascular disorders) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0)
OTHER ADVERSE EVENTS (reported when occurring in more than 5% of participants in an arm); cells are participants affected of the arm's N at risk (number of events):
Term (organ system) | Part A: Dose Escalation (N=20) | Part B: Dose Expansion Cohort (N=29) | Part C: Dose Expansion Cohort (N=13) | Part D: Dose Expansion Cohort (N=12) | Part E: Dose Expansion Cohort (N=17) | Part F: Dose Expansion Cohort (N=20)
Rash (Skin and subcutaneous tissue disorders) | 8 (9) | 23 (26) | 10 (13) | 11 (12) | 16 (17) | 18 (26)
Dry skin (Skin and subcutaneous tissue disorders) | 9 (9) | 14 (14) | 5 (6) | 2 (2) | 5 (5) | 3 (3)
Pruritus (Skin and subcutaneous tissue disorders) | 6 (6) | 13 (14) | 5 (7) | 1 (1) | 7 (8) | 5 (6)
Skin fissures (Skin and subcutaneous tissue disorders) | 4 (6) | 10 (14) | 4 (4) | 2 (4) | 2 (4) | 10 (14)
Erythema (Skin and subcutaneous tissue disorders) | 1 (2) | 7 (8) | 3 (4) | 0 (0) | 2 (2) | 1 (1)
Dermatitis acneiform (Skin and subcutaneous tissue disorders) | 6 (6) | 5 (5) | 0 (0) | 0 (0) | 1 (1) | 2 (2)
Alopecia (Skin and subcutaneous tissue disorders) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 1 (1) | 2 (2)
Eczema (Skin and subcutaneous tissue disorders) | 0 (0) | 2 (2) | 1 (1) | 1 (1) | 0 (0) | 0 (0)
Hypertrichosis (Skin and subcutaneous tissue disorders) | 1 (1) | 3 (3) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Nail toxicity (Skin and subcutaneous tissue disorders) | 0 (0) | 2 (2) | 0 (0) | 0 (0) | 0 (0) | 1 (1)
Onycholysis (Skin and subcutaneous tissue disorders) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 1 (1) | 1 (1)
Pain of skin (Skin and subcutaneous tissue disorders) | 2 (2) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Rash maculo-papular (Skin and subcutaneous tissue disorders) | 3 (3) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Palmar-plantar erythrodysaesthesia syndrome (Skin and subcutaneous tissue disorders) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 1 (1) | 0 (0)
Scab (Skin and subcutaneous tissue disorders) | 0 (0) | 2 (2) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Skin hyperpigmentation (Skin and subcutaneous tissue disorders) | 0 (0) | 1 (1) | 1 (1) | 0 (0) | 0 (0) | 0 (0)
Acne (Skin and subcutaneous tissue disorders) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0)
Skin exfoliation (Skin and subcutaneous tissue disorders) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0)
Rash erythematous (Skin and subcutaneous tissue disorders) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0)
Asthenia (General disorders) | 1 (1) | 7 (11) | 7 (10) | 7 (11) | 7 (10) | 8 (14)
Mucosal inflammation (General disorders) | 6 (8) | 10 (16) | 4 (7) | 1 (6) | 4 (6) | 5 (8)
Xerosis (General disorders) | 0 (0) | 8 (8) | 2 (2) | 1 (1) | 5 (5) | 3 (4)
Edema peripheral (General disorders) | 2 (2) | 4 (4) | 3 (3) | 2 (2) | 0 (0) | 1 (1)
Fatigue (General disorders) | 3 (3) | 4 (4) | 1 (1) | 0 (0) | 0 (0) | 0 (0)
Edema (General disorders) | 2 (2) | 1 (1) | 1 (1) | 1 (2) | 0 (0) | 0 (0)
Chills (General disorders) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 1 (1) | 1 (1)
Device occlusion (General disorders) | 0 (0) | 2 (2) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Pyrexia (General disorders) | 1 (2) | 3 (3) | 0 (0) | 1 (1) | 2 (5) | 7 (10)
Diarrhea (Gastrointestinal disorders) | 6 (9) | 10 (14) | 7 (13) | 4 (7) | 10 (20) | 7 (12)
Nausea (Gastrointestinal disorders) | 3 (5) | 8 (13) | 3 (3) | 4 (4) | 2 (2) | 2 (4)
Vomiting (Gastrointestinal disorders) | 0 (0) | 5 (9) | 4 (8) | 3 (5) | 1 (1) | 2 (5)
Constipation (Gastrointestinal disorders) | 0 (0) | 4 (4) | 2 (4) | 0 (0) | 3 (4) | 4 (6)
Abdominal pain (Gastrointestinal disorders) | 0 (0) | 3 (3) | 0 (0) | 3 (3) | 2 (2) | 2 (4)
Dyspepsia (Gastrointestinal disorders) | 1 (1) | 2 (2) | 1 (1) | 1 (1) | 0 (0) | 0 (0)
Stomatitis (Gastrointestinal disorders) | 0 (0) | 2 (2) | 1 (1) | 0 (0) | 1 (1) | 0 (0)
Abdominal pain upper (Gastrointestinal disorders) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 2 (2)
Ascites (Gastrointestinal disorders) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0)
Hemorrhoids (Gastrointestinal disorders) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0)
Flatulence (Gastrointestinal disorders) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 3 (3)
Dry mouth (Gastrointestinal disorders) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0)
Hypomagnesemia (Metabolism and nutrition disorders) | 5 (5) | 17 (19) | 6 (8) | 7 (9) | 12 (15) | 9 (14)
Decreased appetite (Metabolism and nutrition disorders) | 0 (0) | 9 (9) | 5 (6) | 4 (4) | 2 (2) | 4 (6)
Hypocalcemia (Metabolism and nutrition disorders) | 0 (0) | 10 (11) | 1 (1) | 1 (1) | 1 (1) | 4 (4)
Hypokalemia (Metabolism and nutrition disorders) | 1 (1) | 2 (4) | 3 (3) | 2 (2) | 0 (0) | 2 (2)
Hyperglycemia (Metabolism and nutrition disorders) | 1 (1) | 2 (2) | 1 (1) | 1 (1) | 2 (2) | 1 (1)
Hypophosphatemia (Metabolism and nutrition disorders) | 0 (0) | 2 (2) | 0 (0) | 0 (0) | 0 (0) | 1 (1)
Hyperkalemia (Metabolism and nutrition disorders) | 1 (1) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0)
Hypoalbuminemia (Metabolism and nutrition disorders) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 1 (1) | 0 (0)
Iron deficiency (Metabolism and nutrition disorders) | 0 (0) | 2 (2) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Hypertriglyceridemia (Metabolism and nutrition disorders) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0)
Paronychia (Infections and infestations) | 3 (4) | 9 (15) | 2 (4) | 2 (4) | 4 (5) | 3 (3)
Superinfection (Infections and infestations) | 2 (4) | 6 (8) | 1 (2) | 0 (0) | 0 (0) | 0 (0)
Urinary tract infection (Infections and infestations) | 1 (1) | 1 (2) | 1 (1) | 1 (1) | 2 (2) | 2 (3)
Nasopharyngitis (Infections and infestations) | 0 (0) | 2 (2) | 0 (0) | 0 (0) | 1 (1) | 3 (4)
Respiratory tract infection (Infections and infestations) | 2 (2) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 2 (2)
Gastroenteritis (Infections and infestations) | 1 (1) | 1 (1) | 1 (1) | 0 (0) | 0 (0) | 0 (0)
Skin infection (Infections and infestations) | 1 (1) | 1 (1) | 1 (1) | 0 (0) | 0 (0) | 0 (0)
Upper respiratory tract infection (Infections and infestations) | 2 (4) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Fungal infection (Infections and infestations) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0)
Nail infection (Infections and infestations) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0)
Aspartate aminotransferase increased (Investigations) | 1 (1) | 0 (0) | 0 (0) | 1 (1) | 3 (3) | 3 (4)
Alanine aminotransferase increased (Investigations) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 2 (2) | 3 (4)
Blood alkaline phosphatase increase (Investigations) | 0 (0) | 1 (1) | 0 (0) | 1 (1) | 0 (0) | 2 (2)
Blood magnesium decreased (Investigations) | 1 (1) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 1 (1)
Hemoglobin decreased (Investigations) | 0 (0) | 1 (1) | 0 (0) | 1 (1) | 0 (0) | 0 (0)
Body temperature decreased (Investigations) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0)
Amylase increased (Investigations) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 1 (1)
Blood albumin decreased (Investigations) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 1 (1)
Lipase increased (Investigations) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 1 (1)
Blood creatinine increased (Investigations) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0)
Platelet count decreased (Investigations) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0)
Conjunctivitis (Eye disorders) | 1 (1) | 10 (14) | 2 (4) | 1 (1) | 4 (4) | 1 (2)
Dry eye (Eye disorders) | 1 (1) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 2 (2)
Blepharitis (Eye disorders) | 0 (0) | 1 (1) | 2 (2) | 0 (0) | 0 (0) | 0 (0)
Lacrimation increased (Eye disorders) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0)
Ocular icterus (Eye disorders) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0)
Back pain (Musculoskeletal and connective tissue disorders) | 2 (3) | 1 (1) | 1 (1) | 1 (1) | 1 (1) | 3 (4)
Musculoskeletal pain (Musculoskeletal and connective tissue disorders) | 2 (2) | 1 (2) | 1 (1) | 0 (0) | 0 (0) | 1 (1)
Muscle spasms (Musculoskeletal and connective tissue disorders) | 1 (1) | 1 (1) | 1 (1) | 0 (0) | 0 (0) | 0 (0)
Arthralgia (Musculoskeletal and connective tissue disorders) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 1 (1)
Bone pain (Musculoskeletal and connective tissue disorders) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0)
Groin pain (Musculoskeletal and connective tissue disorders) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0)
Musculoskeletal stiffness (Musculoskeletal and connective tissue disorders) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0)
Dyspnea (Respiratory, thoracic and mediastinal disorders) | 3 (3) | 5 (5) | 3 (3) | 0 (0) | 0 (0) | 1 (1)
Cough (Respiratory, thoracic and mediastinal disorders) | 2 (2) | 3 (3) | 1 (1) | 1 (1) | 0 (0) | 0 (0)
Productive cough (Respiratory, thoracic and mediastinal disorders) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 2 (2)
Wheezing (Respiratory, thoracic and mediastinal disorders) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0)
Headache (Nervous system disorders) | 2 (2) | 0 (0) | 1 (1) | 1 (1) | 2 (5) | 0 (0)
Dysgeusia (Nervous system disorders) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 3 (3) | 1 (1)
Neuropathy peripheral (Nervous system disorders) | 1 (1) | 1 (1) | 0 (0) | 1 (1) | 0 (0) | 0 (0)
Infusion related reaction (Injury, poisoning and procedural complications) | 3 (3) | 1 (2) | 0 (0) | 1 (1) | 2 (4) | 2 (3)
Procedural pain (Injury, poisoning and procedural complications) | 0 (0) | 2 (2) | 1 (1) | 0 (0) | 0 (0) | 0 (0)
Ligament sprain (Injury, poisoning and procedural complications) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0)
Toxicity to various agents (Injury, poisoning and procedural complications) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0)
Anemia (Blood and lymphatic system disorders) | 1 (1) | 4 (4) | 0 (0) | 1 (1) | 3 (3) | 2 (2)
Thrombocytopenia (Blood and lymphatic system disorders) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 1 (1) | 0 (0)
Leukocytosis (Blood and lymphatic system disorders) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0)
Hyperbilirubinemia (Hepatobiliary disorders) | 0 (0) | 1 (1) | 1 (1) | 1 (1) | 2 (2) | 1 (1)
Hepatic pain (Hepatobiliary disorders) | 1 (1) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 2 (2)
Insomnia (Psychiatric disorders) | 0 (0) | 3 (3) | 0 (0) | 0 (0) | 0 (0) | 2 (2)
Depression (Psychiatric disorders) | 0 (0) | 1 (1) | 1 (1) | 0 (0) | 0 (0) | 0 (0)
Anxiety (Psychiatric disorders) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0)
Tumor pain (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 1 (2) | 0 (0) | 1 (1) | 0 (0) | 1 (1) | 0 (0)
Tumor associated fever (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0)
Hypersensitivity (Immune system disorders) | 1 (11) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 1 (1)
Hypertension (Vascular disorders) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 1 (1) | 0 (0)
Trichomegaly (Congenital, familial and genetic disorders) | 0 (0) | 2 (2) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Metrorrhagia (Reproductive system and breast disorders) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 2 (2)
Atrophic vulvovaginitis (Reproductive system and breast disorders) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0)
Pruritus genital (Reproductive system and breast disorders) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0)
Dysuria (Renal and urinary disorders) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0)
Leukocyturia (Renal and urinary disorders) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0)
Urinary incontinence (Renal and urinary disorders) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0)

LIMITATIONS AND CAVEATS:
None reported

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: No; Agreement restricts PI disclosure of results: No